CLINICAL TRIAL: NCT06075329
Title: Dementia Caregivers and Contemplative Practice: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Nirmala Lekhak, PhD, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2023-395
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contemplative Practice (Experimental): Maitribodh Sambodh (MSD) is a unique form of contemplative practice which combines breath watch, mantra or vibrational sound chant, focused meditation followed by loving kindness or a gratitude exercise at the end.
  Interventions: Behavioral: Contemplative Practice
- Waitlist Control (Other): The arm will eventually get the intervention.
  Interventions: Behavioral: Contemplative Practice

INTERVENTIONS:
Behavioral: Contemplative Practice — Contemplative practice included Maitribodh Sambodh Dhyaan (MSD), which was designed to increase feeling of love and connection by including most of components of different contemplative practices such as breath watch, mantra or vibrational sound chant, focused meditation, and visualization followed by loving-kindness or a gratitude exercise at the end.

SUMMARY:
The goal of this study is to test the contemplative practice is feasible and acceptable among informal dementia caregivers population at all stages.

DETAILED DESCRIPTION:
It will also examine the benefits of this intervention and compare the outcomes between two groups (intervention and wait-list control).

ELIGIBILITY:
Inclusion Criteria:

* Dementia Family Caregivers
* At least cared for dementia care receipient more than 6 months

Exclusion Criteria:

* If they have meditated less than 2 months ago
* Cognitive or language barrier that would make it difficult to understand and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Loneliness | baseline, at 10 days and 21 days of Matribodh Sambodh Dhyaan practice (meditation), and at 30 days and 60 days follow-up.
  The UCLA 3-item Loneliness scale will be used to measure loneliness. The scores on this scale range from 3 to 9, the highest scores indicative of a higher level of loneliness. The scale is called UCLA 3-item scale but UCLA is representative of University of California Los Angeles.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmala Lekhak, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No